CLINICAL TRIAL: NCT04387877
Title: The Effect of Graston Technique in Deep Gluteal Syndrome
Brief Title: Graston Technique in Deep Gluteal Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019.308.IRB1.052
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-02

CONDITIONS: Deep Gluteal Syndrome; Piriformis Syndrome
Keywords: deep gluteal syndrome; graston; elastography; piriformis syndrome; miyofascial release
MeSH Terms: conditions — Hip socket neuropathy; Piriformis Muscle Syndrome | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graston Group (Experimental): Graston technique will be applied on the lateral and posterior myofascial chain area tensor fascia lata, gluteus medius, gluteus minimus, gluteus maximus, hamstring, gastrocnemius and soleus muscles) in 15 minutes.
  Interventions: Device: Graston
- Sham Group (Sham Comparator): Sham graston technique will be applied on lateral and posterior myofascial chain area (tensor fascia lata, gluteus medius, gluteus minimus, gluteus maximus, hamstring, gastrocnemius and soleus muscles) in 15 minutes.
  (Sham graston technique will be applied to the patient by partially touching the muscle or fascia region via ultrasound gel with the flat part of the Graston tool so as not to provide the activity of the fascia)
  Interventions: Other: Sham

INTERVENTIONS:
Device: Graston — Graston technique will be applied on the lateral and posterior fascia (tensor fascia lata, gluteus medius, gluteus minimus, gluteus maximus, hamstring, gastrocnemius and soleus muscles) in 15 minutes.
  For the first 2 weeks; dorsolumbar stabilization, straight and side leg lifting, gluteal setting, side walking exercises For the second 2 weeks; dorsolumbar stabilization counting on spot, straight and side leg lifting, gluteal setting, side walking exercises with 0.5 kg weight on the ankle, piriformis, tensor fascia lata and hamstring stretching exercises
  Arms: Graston Group
Other: Sham — Sham graston technique will be applied on lateral and posterior fascia (tensor fascia lata, gluteus medius, gluteus minimus, gluteus maximus, hamstring, gastrocnemius and soleus muscles) in 15 minutes.
  (Sham graston technique will be applied by partially touching the skin overlying the muscle or fascia region via ultrasound gel with the flat part of the Graston instrument so as not to provide any activity of the fascia) For the first 2 weeks; dorsolumbar stabilization, counting on spot, straight and side leg lifting, gluteal setting, side walking exercises For the second 2 weeks; dorsolumbar stabilization counting on spot, straight and side leg lifting, gluteal setting, side walking exercises with 0.5 kg weight on the ankle, piriformis, tensor fascia lata and hamstring stretching exercises
  Arms: Sham Group

SUMMARY:
Deep gluteal syndrome describes the presence of pain in the buttock caused from non-discogenic and extrapelvic entrapment of the sciatic nerve. The Graston Technique (GT) is a kind of manual therapy technique known as soft-tissue instrument-assisted mobilization. Instruments help to perform massage/scraping of the skin and miyofascia gently. The aim of this study is to investigate additive effect of GT applied to the lateral and posterior fascia to the exercise program in patients with deep gluteal syndrome on pain and disability.

DETAILED DESCRIPTION:
Deep gluteal syndrome describes the presence of pain in the buttock caused from non-discogenic and extrapelvic entrapment of the sciatic nerve. Several structures can be involved in sciatic nerve entrapment within the gluteal space [1]. There are many anatomical variations between the sciatic nerve and piriformis muscle (PM) [2]. Some authors have associated deep gluteal pain syndrome with piriformis syndrome (PS) [3]. Chronic buttock pain caused by the musculoskeletal pathologies of the PM such as myofascial pain or pinching of the sciatic nerve by the PM during certain leg and hip maneuvers [4]. In most cases, PS is widely believed to be myofascial in origin [5].

Treatment of PS starts with conservative pharmacotherapy with nonsteroidal anti-inflammatory drugs, muscle relaxants, and neuropathic pain agents and continues with physical therapy, which includes stretching of the PM to correct the underlying pathology [6]. If the conservative regimen fails, then more aggressive therapy, such as local injection of PM, which may reconfirm the diagnosis through therapeutic success, should be performed [7].

Myofascial release is a specific manual therapy method claimed to be useful for treating skeletal muscle immobility and pain by relaxing contracted muscles, improving blood, oxygen, and lymphatic circulation, and stimulating the stretch reflex in muscles [8]. The Graston Technique (GT) is a form of manual therapy known as soft-tissue instrument-assisted mobilization. It is one of a number of manual therapy approaches that uses instruments with a specialized form of massage/scraping the skin and miyofascia gently [9]. This technique seems to have the therapeutic effects of inhibiting the adhesion of tissue, increasing the number of fibroblasts, and promoting collagen synthesis [10].

Gait analysis has been widely used in the diagnosis of locomotors pathology and the assessment of treatment. But study of gait on deep gluteal syndrome remain unclear. 3-D motion analysis can be used to measure the kinematic and kinetic together with temporal-spatial parameters data of patients with deep gluteal syndrome during walking. Patients with deep gluteal syndrome show significant increase gait speed and cadence, and peak extensor moments with increased flexion, abduction and internal rotation at the hip during the whole gait cycle [11].

Shear Wave elastography is an imaging technique which quantifies tissue stiffness by measuring the speed of shear waves in tissue. It is a new advanced dynamic ultrasound technique that provides information about the stiffness / consistency of the tissue by measuring the degree of strain in the tissue without external force [12].

The aim of this study is to investigate the additive effect of GT to the exercise program in patients with deep gluteal syndrome on pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 70
* Having unilateral hip and/or leg pain with positive FAIR (flexion, adduction, internal rotation) test
* Tenderness and/or trigger point at the Piriformis with deep palpation

Exclusion Criteria:

* Neurological deficit
* Limited lumbar and/or hip range of motion
* Previous surgery of the lumbar and/ or hip region
* Being in gestational or lactational period
* Body mass index greater than 35
* Inflammatory or infectious disease
* Active psychiatric disease
* Uncontrolled hypertension
* Uncontrolled diabetes mellitus
* Noncompensated chronic heart/liver/renal deficiency or vascular/tumoral disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 4 weeks
  Oswestry Disability Index (ODI), measures the level of disability. It consists of 10 items questioning the severity of pain, self-care, lifting and carrying, walking, sitting, standing, sleep, the degree of pain change, travel and social life. Its Turkish version is validated in 2004. Items are scored between 0 and 5, and the total score is multiplied by two. The maximum score is "100". As the total score increases, the level of disability increases.

SECONDARY OUTCOMES:
Visual Analog Scale | 4 weeks
  It is a scale consisting of a 10-centimeter line that evaluates the intensity of pain. Starting point of scale, 0 = no pain, end point 10 = expressed as the most severe pain encountered in life. Patients are asked to mark the severity of pain on the line. When calculating, the distance between the marked point and the starting point is measured in centimeters. Increasing the score means that the pain intensity increases.
Nottingham Health Profile | 4 weeks
  Nottingham health profile is a general quality-of-life questionnaire that measures health problems that a person perceives and how these problems affect normal and daily activities. The questionnaire consists of 38 items and evaluates 6 dimensions related to health: energy, pain, emotional reactions, sleep, social isolation and physical activity. Questions are answered as yes or no. Scoring is done in every section between 0-100. 0 indicates the best health status, 100 worst health status. The total Nottingham Health Profile score is obtained from the sum of the sub-scores. Turkish validity and reliability were shown in 2000.
Shearwave Elastography | 4 weeks
  Thickness and shear wave elastography (SWE) of tensor fascia lata (TFL), proximal and distal part of iliotibial band (ITB) on the affected side of the body in side lying position were evaluated at rest using GE LOGIQ E9 XDclear ultrasound device equipped with lineer array transducer (9L-D, B-mode, frequency 9-5 MHz). We measured shear wave velocity (SWV) (expressed in m/s) and young modulus (in kPa). Three 5 mm diameter region of interest (ROI) was located most homogeneous part of the color map. For sufficient image quality and shear wave signals a large amount of gel was used and minimum pressure was applied on the probe. The positions of transducers were selected after browsing previous studies and testing on different subjects. The same specialist performed all the evaluation on the same subjects before and after treatment.
Gait Analyze | 4 weeks
  The Noraxon myoMOTION™ software module features a medically accurate avatar paired with a toolset for analyzing pre-processed motion records. Real-time data is automatically synchronized in an all-in-one analysis. In our study, each subject is stick with 13 retroreflective markers on the bony landmarks for tracking the motions of the body segments, including the head, each superor iliac spine, each middle of humerus, each wrist, each metacarp, head of fibula, each navicular tuberosity. By using the 1-cameras motion analysis system (The Noraxon myoMOTION™) and measuring the ground reaction forces with a forceplate (The Noraxon myoPressure™)

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozyemisci Taskiran, Prof, Principal Investigator — Koc University School of Medicine
Locations (1):
- Koc University School of Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Martin HD, Reddy M, Gomez-Hoyos J. Deep gluteal syndrome. J Hip Preserv Surg. 2015 Jul;2(2):99-107. doi: 10.1093/jhps/hnv029. Epub 2015 Jun 6. PMID 27011826
- [Result] Natsis K, Totlis T, Konstantinidis GA, Paraskevas G, Piagkou M, Koebke J. Anatomical variations between the sciatic nerve and the piriformis muscle: a contribution to surgical anatomy in piriformis syndrome. Surg Radiol Anat. 2014 Apr;36(3):273-80. doi: 10.1007/s00276-013-1180-7. Epub 2013 Jul 31. PMID 23900507
- [Result] Carro LP, Hernando MF, Cerezal L, Navarro IS, Fernandez AA, Castillo AO. Deep gluteal space problems: piriformis syndrome, ischiofemoral impingement and sciatic nerve release. Muscles Ligaments Tendons J. 2016 Dec 21;6(3):384-396. doi: 10.11138/mltj/2016.6.3.384. eCollection 2016 Jul-Sep. PMID 28066745
- [Result] Santamato A, Micello MF, Valeno G, Beatrice R, Cinone N, Baricich A, Picelli A, Panza F, Logroscino G, Fiore P, Ranieri M. Ultrasound-Guided Injection of Botulinum Toxin Type A for Piriformis Muscle Syndrome: A Case Report and Review of the Literature. Toxins (Basel). 2015 Aug 10;7(8):3045-56. doi: 10.3390/toxins7083045. PMID 26266421
- [Result] Shah JP, Thaker N, Heimur J, Aredo JV, Sikdar S, Gerber L. Myofascial Trigger Points Then and Now: A Historical and Scientific Perspective. PM R. 2015 Jul;7(7):746-761. doi: 10.1016/j.pmrj.2015.01.024. Epub 2015 Feb 24. PMID 25724849
- [Result] Han SK, Kim YS, Kim TH, Kang SH. Surgical Treatment of Piriformis Syndrome. Clin Orthop Surg. 2017 Jun;9(2):136-144. doi: 10.4055/cios.2017.9.2.136. Epub 2017 May 8. PMID 28567214
- [Result] Misirlioglu TO, Akgun K, Palamar D, Erden MG, Erbilir T. Piriformis syndrome: comparison of the effectiveness of local anesthetic and corticosteroid injections: a double-blinded, randomized controlled study. Pain Physician. 2015 Mar-Apr;18(2):163-71. PMID 25794202
- [Result] McKenney K, Elder AS, Elder C, Hutchins A. Myofascial release as a treatment for orthopaedic conditions: a systematic review. J Athl Train. 2013 Jul-Aug;48(4):522-7. doi: 10.4085/1062-6050-48.3.17. Epub 2013 Apr 3. PMID 23725488
- [Result] Looney B, Srokose T, Fernandez-de-las-Penas C, Cleland JA. Graston instrument soft tissue mobilization and home stretching for the management of plantar heel pain: a case series. J Manipulative Physiol Ther. 2011 Feb;34(2):138-42. doi: 10.1016/j.jmpt.2010.12.003. PMID 21334547
- [Result] Moon JH, Jung JH, Won YS, Cho HY. Immediate effects of Graston Technique on hamstring muscle extensibility and pain intensity in patients with nonspecific low back pain. J Phys Ther Sci. 2017 Feb;29(2):224-227. doi: 10.1589/jpts.29.224. Epub 2017 Feb 24. PMID 28265144
- [Result] Huang, H.P., et al., Gait Analysis of Patients with Unilateral Piriformis Syndrome. IFMBE Proceedings, 2015. 47: p. 104-106.
- [Result] Sarvazyan A, Hall TJ, Urban MW, Fatemi M, Aglyamov SR, Garra BS. AN OVERVIEW OF ELASTOGRAPHY - AN EMERGING BRANCH OF MEDICAL IMAGING. Curr Med Imaging Rev. 2011 Nov;7(4):255-282. doi: 10.2174/157340511798038684. PMID 22308105
- [Result] Creze M, Nordez A, Soubeyrand M, Rocher L, Maitre X, Bellin MF. Shear wave sonoelastography of skeletal muscle: basic principles, biomechanical concepts, clinical applications, and future perspectives. Skeletal Radiol. 2018 Apr;47(4):457-471. doi: 10.1007/s00256-017-2843-y. Epub 2017 Dec 9. PMID 29224123
- [Result] Deshmukh S, Abboud SF, Grant T, Omar IM. High-resolution ultrasound of the fascia lata iliac crest attachment: anatomy, pathology, and image-guided treatment. Skeletal Radiol. 2019 Sep;48(9):1315-1321. doi: 10.1007/s00256-018-3141-z. Epub 2019 Jan 7. PMID 30617717
- [Result] Whittaker JL, Emery CA. Sonographic measures of the gluteus medius, gluteus minimus, and vastus medialis muscles. J Orthop Sports Phys Ther. 2014 Aug;44(8):627-32. doi: 10.2519/jospt.2014.5315. Epub 2014 Jul 16. PMID 25029916